CLINICAL TRIAL: NCT06314178
Title: Assessing Demographic Biases in Deep Learning Model for Fetal Growth Estimation in Clinical Practice
Brief Title: Assessing Demographic Biases in Deep Learning Model for Fetal Growth Estimation in Clinical Practice. Patients Eligible for Inclusion Are Women with a Gestational Age Between 24-42 Weeks Undergoing a Third-trimester Growth Scan. the Image Data from the Scan Are Used to Calculate Fetal Weight.
Status: Completed | Type: Observational
Sponsor: Copenhagen Academy for Medical Education and Simulation (Other)
Responsible Party: Principal Investigator, Julie Leth-Petersen, Principal Investigator, Copenhagen Academy for Medical Education and Simulation
Other Study IDs: p-2024-15469
Record Dates: First submitted 2024-03-06; First posted 2024-03-15 (Actual); Last update posted 2024-12-04 (Actual); Status verified 2024-12

CONDITIONS: Pregnancy Complications
MeSH Terms: conditions — Pregnancy Complications

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

GROUPS / COHORTS (1):
- Pregnant women between 24-42 weeks of gestation: No interventions

SUMMARY:
The goal of this observational study is to compare a new artificial intelligence (AI) feedback tool with the traditional method for estimating fetal weight during ultrasound scans on pregnant women between 24-42 weeks of gestation. The study aims to investigate the presence of demographic bias in the AI model. The demographic factors examined in the study include Body Mass Index (BMI), the number of births, fetal age, mother's age, fetal sex, and the presence of preeclampsia. Moreover, the study will compare the accuracy of the AI model and the Hadlock model, a fetal growth formula, in estimating fetal weight. Participants will have their ultrasound scans pseudonymized and securely stored on password-protected removable drives, ensuring their identity and privacy are maintained. Afterward, the ultrasound data will be sent to the Technical University of Denmark (DTU), where the AI model will analyze the images to estimate fetal weight.

ELIGIBILITY:
Inclusion Criteria:

* Women with gestational age between 24-42 weeks undergoing a third-trimester growth scan.

Exclusion Criteria:

* Women with multiple pregnancies.

Sex: Female | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Gender Based: Yes — Pregnant women between 24-42 weeks of gestation.
Study Population: Department of Prenatal Examinations at Rigshospitalet, Copenhagen, Denmark.
Sampling Method: Non-Probability Sample
Enrollment: 185 (Actual)
Dates: Start 2024-07-01 (Actual); Primary Completion 2024-08-30 (Actual); Study Completion 2024-11-30 (Actual)

PRIMARY OUTCOMES:
Demographic biases | From enrollment to the birth of the child
  The primary objective is to investigate potential demographic biases inherent in the deep learning model developed for estimating fetal growth in clinical practice. This is achieved by comparing the relative error between fetal weight at scan time (this value is extrapolated from the birth weight using the Marsal growth curve) and estimations from the Hadlock formula and the deep learning model.

SECONDARY OUTCOMES:
Comparing the accuracy of the Hadlock formula and the AI model | From enrollment to the birth of the child
  The secondary objective is to compare the accuracy of fetal weight estimation between the Hadlock formula and a deep learning model in clinical practice using a paired t-test.

CONTACTS AND LOCATIONS:
Locations (1):
- Copenhagen University Hospital, Rigshospitalet, Copenhagen, Denmark

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Background] Salomon LJ, Alfirevic Z, Da Silva Costa F, Deter RL, Figueras F, Ghi T, Glanc P, Khalil A, Lee W, Napolitano R, Papageorghiou A, Sotiriadis A, Stirnemann J, Toi A, Yeo G. ISUOG Practice Guidelines: ultrasound assessment of fetal biometry and growth. Ultrasound Obstet Gynecol. 2019 Jun;53(6):715-723. doi: 10.1002/uog.20272. PMID 31169958